CLINICAL TRIAL: NCT02848027
Title: Correlating the Osteoarthritic Knee Microenvironment to Clinical Outcome After Treatment With Regenexx®SD Treatment
Acronym: KneeOA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Regenexx, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RSI2015-LAB02
Record Dates: First submitted 2015-09-30; First posted 2016-07-28 (Estimated); Last update posted 2022-07-08 (Actual); Status verified 2022-07

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Regenexx-SD procedure (Experimental): Measure components of knee synovial fluid collected 2-4 days before and after Regenexx SD procedure
  Interventions: Biological: Regenexx SD® procedure

INTERVENTIONS:
Biological: Regenexx SD® procedure — Correlate patient outcomes 6 months after receiving the Regenexx SD procedure with measurements of synovial fluid collected before and after procedure.

SUMMARY:
Single-center, lab blinded to include up to 400 subjects with knee osteoarthritis. Collection of synovial fluid from diseased knee before and after Regenexx®SD treatment will serve as the experimental condition, i.e. the osteoarthritic knee.

DETAILED DESCRIPTION:
Single-center, laboratory blinded to include up to 400 subjects with knee osteoarthritis in unilateral or bilateral knees treated with Regenexx® SD in the osteoarthritic knee/s.Initial study procedures include baseline evaluation of medical history, knee history, knee examination, medication use, MRI, and subject-reported outcomes.

Subjects will be enrolled within the 120 days prior to Regenexx® SD injection. A preoperative visit will occur at the time of enrollment. Collection of synovial fluid from the OA knee/s will serve as the experimental condition, i.e. the osteoarthritic knee.Each osteoarthritic subject will undergo withdrawal of knee joint synovial fluid for each knee being treated (0.3-0.5 ml) which will be analyzed by the research laboratory via multiplexed enzyme linked immunosorbent assay (ELISA) and dimethylmethylene blue assay (DMMB) at pre-injection (2-8 days before Regenexx® SD treatment) and post-injection (2-8 days after Regenexx® SD). Documentation of osteoarthritic joint characteristics and injection procedure details will be recorded throughout the study.

The unaffected knee joint will undergo no treatment, but bilateral knees may be treated.

Components of the synovial fluid will be correlated to post-treatment clinical outcomes, which include patient-reported questionnaires as well as assessment of post-injection complications, adverse events, re-injections and surgical interventions. Patient-reported clinical outcomes are comprised of the IKDC Subjective Knee Evaluation, the Lower Extremity Function Scale, Numeric Pain Scale and a Patient Reported Percent Improvement form.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary signature of the IRB approved Informed Consent
2. Unilateral or bilateral osteoarthritic male or female ages 35-85
3. Pain, swelling, and/or functional disability in the affected knee consistent with osteoarthritis in the knee joint
4. Physical examination consistent with osteoarthritis in one knee joint
5. Kellgren-Lawrence grade 2 or greater knee osteoarthritis and/or diagnostic MRI imaging of the affected knee showing osteoarthritis (i.e. chondral loss, fissuring, defect, bone marrow lesion, meniscus tear, synovial thickening, etc…)
6. Is independent, ambulatory, and can comply with all post-operative evaluations and visits

Exclusion Criteria:

1. Knee injections of any type within 3 months prior to the study.
2. Knee surgery within 6 months prior to the study.
3. Inflammatory or auto-immune based joint diseases or other lower extremity pathology (e.g., rheumatoid arthritis, systemic lupus erythematosus, psoriatic arthritis, polymyalgia, polymyositis, gout pseudogout)
4. Quinolone or Statin induced myopathy/tendinopathy
5. Severe neurogenic inflammation of the cutaneous nerves about the knee or thigh
6. Contraindications for MRI
7. Condition represents a worker's compensation case
8. Currently involved in a health-related litigation procedure
9. Is pregnant
10. Bleeding disorders
11. Currently taking anticoagulant or immunosuppressive medication
12. Allergy or intolerance to study medication
13. Use of chronic opioid
14. Documented history of drug abuse within six months of treatment
15. Any other condition, that in the opinion of the investigator, that would preclude the patient from enrollment

Ages: 35 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2015-09-08 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2021-08-19 (Actual)

PRIMARY OUTCOMES:
Correlation between components in knee synovial fluid to patient-reported outcomes post-procedure. | 6 months after Regenexx-SD procedure
  Synovial fluid components include cytokine, matrix metalloproteinase levels, and catabolic cartilage breakdown products. These components of synovial fluid will be correlated to the following patient-reported outcomes 6 months after procedure: the International Knee Documentation Committee (IKDC) Subjective Knee Evaluation form.

SECONDARY OUTCOMES:
Comparison of synovial fluid contents | fluid taken ~2-4 days before procedure and ~2-4 days after procedure
  Comparison of cytokine, matrix metalloproteinase concentration levels and cartilage breakdown product levels from pre-Regenexx SD treatment to post-Regenexx SD treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Neven Steinmetz, Ph.D., Study Director — Regenexx, LLC; Christopher J Centeno, M.D., Principal Investigator — Regenexx, LLC

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bain BJ. Morbidity associated with bone marrow aspiration and trephine biopsy - a review of UK data for 2004. Haematologica. 2006 Sep;91(9):1293-4. PMID 16956842
- [Background] Centeno CJ, Schultz JR, Cheever M, Freeman M, Faulkner S, Robinson B, Hanson R. Safety and complications reporting update on the re-implantation of culture-expanded mesenchymal stem cells using autologous platelet lysate technique. Curr Stem Cell Res Ther. 2011 Dec;6(4):368-78. doi: 10.2174/157488811797904371. PMID 22023622
- [Background] Centeno CJ, Schultz JR, Cheever M, Robinson B, Freeman M, Marasco W. Safety and complications reporting on the re-implantation of culture-expanded mesenchymal stem cells using autologous platelet lysate technique. Curr Stem Cell Res Ther. 2010 Mar;5(1):81-93. doi: 10.2174/157488810790442796. PMID 19951252
- [Background] Nejadnik H, Hui JH, Feng Choong EP, Tai BC, Lee EH. Autologous bone marrow-derived mesenchymal stem cells versus autologous chondrocyte implantation: an observational cohort study. Am J Sports Med. 2010 Jun;38(6):1110-6. doi: 10.1177/0363546509359067. Epub 2010 Apr 14. PMID 20392971
- [Background] Wakitani S, Okabe T, Horibe S, Mitsuoka T, Saito M, Koyama T, Nawata M, Tensho K, Kato H, Uematsu K, Kuroda R, Kurosaka M, Yoshiya S, Hattori K, Ohgushi H. Safety of autologous bone marrow-derived mesenchymal stem cell transplantation for cartilage repair in 41 patients with 45 joints followed for up to 11 years and 5 months. J Tissue Eng Regen Med. 2011 Feb;5(2):146-50. doi: 10.1002/term.299. PMID 20603892
- [Background] Irrgang JJ, Anderson AF, Boland AL, Harner CD, Neyret P, Richmond JC, Shelbourne KD; International Knee Documentation Committee. Responsiveness of the International Knee Documentation Committee Subjective Knee Form. Am J Sports Med. 2006 Oct;34(10):1567-73. doi: 10.1177/0363546506288855. Epub 2006 Jul 26. PMID 16870824